CLINICAL TRIAL: NCT04745377
Title: Mapping the Responses to COVID-19 Vaccination in Patients With Cancer - the ReCOVer Study
Brief Title: Responses to COVID-19 Vaccination in Patients With Cancer
Acronym: ReCOVer
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE_42C/21 ReCOVer study
Record Dates: First submitted 2021-01-15; First posted 2021-02-09 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Cancer
Keywords: COVID-19 vaccination; Cancer patients; Immunity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum for neutralising IgG antibody titers against S1 and S2 proteins of SARS-COV-2 virus
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Healthy volunteers from hospital personnel vaccinated for covid-19, who sign informed consent for recording of outcomes and monitor of antibody titers in 3 timepoints
  Interventions: Diagnostic Test: IgG neutralising antibody titers to S1 and S2 proteins of SARS-COV-2 virus
- Cancer patients: Cancer patients with solid tumours, with active disease and/or undergoing active systemic treatment, who will be vaccinated for covid-19
  Interventions: Diagnostic Test: IgG neutralising antibody titers to S1 and S2 proteins of SARS-COV-2 virus

INTERVENTIONS:
Diagnostic Test: IgG neutralising antibody titers to S1 and S2 proteins of SARS-COV-2 virus — IgG neutralising antibody titers to S1 and S2 proteins of SARS-COV-2 virus

SUMMARY:
This is an observational study that will prospectively record and monitor responses and clinical outcomes of patients with cancer after covid-19 vaccination, including measurements of antibody titers in serum and also record potential factors that affect immunity, such as type and stage of cancer, type and time of systemic therapy in relation to covid-19 vaccination.

DETAILED DESCRIPTION:
It is well recognised that patients with cancer are at an increased risk of severe COVID-19 disease and should be at high prioritisation for vaccination against SARS-CoV-2. In Greece the vaccination of healthcare workers has been initiated in January 2021, elderly citizens as well and for cancer patients of all ages will be initiated early February 2021. There are very little available data on the efficacy of immunisation with vaccines overall in cancer patients, with most existing data involving the influenza vaccine. The covid-19 vaccine trials have not included cancer patients, therefore, the efficacy and duration of immunity in patients with cancer are still unknown. Those patients are often immunocompromised due to their disease or the side-effects of their treatment.

Based on the above this study was designed to prospectively record and monitor patients with cancer after covid-19 vaccination. The study will record and measure clinical outcomes, such as possible infection from covid-19 despite vaccination, severity and mortality, but also possible side effects post vaccination. Within the study serological responses (IgG antibody titers) will also be monitored in three timepoints (prior to vaccination, one month and three months after completion of the two doses of vaccination). Potential factors that affect immunity, will be recorded, such as type and stage of cancer, type and time of systemic therapy in relation to covid-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumours and potentially immunocompromised, ie. currently with active disease and/or undergoing active antineoplastic therapy of any type (chemotherapy, immunotherapy, biologic therapy, targeted therapy) that will be vaccinated for covid-19 within the National Program of Vaccination
* patients must sign informed consent for their data monitoring and also for serum antibody titers to covid-19 vaccination measured in three timepoints, prior to 1st dose and 1 and 3 months post completion of two doses

Exclusion Criteria:

* patients with haematological malignancies are excluded
* patients with prior diagnosis of cancer and now on follow-up without active disease are excluded
* patients on adjuvant hormonal therapy are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumours and potentially immunocompromised, ie. currently with active disease and/or undergoing active antineoplastic therapy of any type (chemotherapy, immunotherapy, biologic therapy, targeted therapy) that will be vaccinated for covid-19 within the National Program of Vaccination.
  Also a group of healthy volunteers from the hospital personnel that have been vaccinated within the National Program of Vaccination and signed informed consent for 3 measurements of antibody titers in serum, at the timepoints described aboved.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Clinical outcome post vaccination | 12 months
  The primary outcome is the rate of COVID-19 infections post vaccination in cancer patients compared to individuals without cancer, measured as confirmed COVID-19 infections by positive PCR COVID-tests (in asymptomatic or symptomatic cases within a period of up to 12 months post vaccination)
Serological outcome post vaccination, immune response to vaccination against COVID-19 (measured as antibody titre 1 month after completion of vaccination | 1 month
  This primary outcome includes the antibody based immune response to COVID-19 vaccination measured 1 month after the complete vaccination (2 doses) in patients with cancer as compared to individuals without cancer, expressed as antibody titres by means of ELISA
Serological outcome post vaccination, immune response to vaccination against COVID-19 (measured as antibody titre 3 months after completion of vaccination | 3 months
  This outcome involves the persistence of antibody response to COVID-19 vaccination measured 3 months after the complete vaccination (2 doses) in patients with cancer as compared to individuals without cancer, expressed as antibody titres by means of ELISA

SECONDARY OUTCOMES:
Safety and Tolerance assessment - AEs; Incidence and severity of Adverse Events post vaccination | 12 months
  Incidence and severity of AEs post vaccination, with incidence and nature of AEs reported after each vaccination dose and up to 12 months post vaccination. The number of participants with adverse events and the severity of adverse events will be recorded as assessed by CTCAE v4.0.
Correlation of factors that might affect immune response in patients with cancer compared to individuals without cancer | 12 months
  Correlation of factors (such as level of White Blood Count and Neutrophil Count prior to vaccination, type of cancer, type of cancer treatment, age and comorbidities) to the level of antibody response mounted post vaccination in patients with cancer. Age-adjusted comparisons with the group of individuals without cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Metropolitan Hospital, Athens, Attica, Greece